CLINICAL TRIAL: NCT00269360
Title: Manipulation, Exercise, and Self-Care for Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Berman Center for Outcomes and Clinical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP10013
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Neck Pain
Keywords: Chiropractic; Manual Therapies; Exercise; Randomized; Clinical Trial; Neck Pain
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Procedure: Chiropractic + Supervised Rehabilitative Exercise
- 2 (Experimental)
  Interventions: Procedure: Supervised Rehabilitative Exercise
- 3 (Active Comparator)
  Interventions: Behavioral: Self-care education

INTERVENTIONS:
Procedure: Chiropractic + Supervised Rehabilitative Exercise — Chiropractic care will include manual spinal manipulation, with light soft tissue massage as indicated to facilitate the spinal manipulative therapy. The spinal levels treated will be determined by the individual chiropractors by static and/or motion palpation.
  Patients will attend 20, 1 hour sessions of rehabilitative exercises for the neck and upper body. Each session will begin with a 10-minute aerobic warm-up of the upper body and five minutes of light stretching to prepare for the strengthening exercises.
  Arms: 1
Procedure: Supervised Rehabilitative Exercise — Patients will attend 20, 1 hour sessions of rehabilitative exercises for the neck and upper body. Each session will begin with a 10-minute aerobic warm-up of the upper body and five minutes of light stretching to prepare for the strengthening exercises.
  Arms: 2
Behavioral: Self-care education — Self-care education will be provided by the therapist trained in the study protocol. Two, one-hour sessions will be given regarding self-care measures and ergonomics relative to work and activities of daily living. These will include postural instructions and practical demonstrations of proper body mechanics performed with patient participation.
  Arms: 3

SUMMARY:
The purpose of this study is to compare three treatments for neck pain: 1) rehabilitative exercise, 2) chiropractic spinal manipulation combined with rehabilitative exercise, and 3) self-care education.

DETAILED DESCRIPTION:
Neck pain is very common, afflicting 10% of the population at any given time. Despite its significant socioeconomic impact, neck pain has been poorly investigated. The broad, long term objective of this interdisciplinary research is to identify effective therapies for neck pain and to increase our knowledge of this problematic condition. This multidisciplinary, randomized clinical trial is based on the investigators' previous neck pain research and will assess three treatment approaches for chronic neck pain:

1. rehabilitative exercise
2. chiropractic spinal manipulation combined with rehabilitative exercise
3. self-care education (a minimal intervention control)

The primary aim of this study is to examine the relative efficacy of the three interventions in terms of patient-rated outcomes in the short term (after 12 weeks) and long term (after 52 weeks) for chronic neck pain. Secondary aims are to assess the relative cost-effectiveness and cost utility of the three treatments, evaluate changes in objective cervical spine function, assess if cervical function is associated with changes in patient-rated outcomes, identify predictors of outcome and finally, to describe patients' interpretations of outcome measures used in clinical trials.

Using previously demonstrated recruitment methods, 270 participants with chronic neck pain will be recruited. Self-reported outcome measures will be collected at baseline and 4, 12, 26 and 52 weeks; objective outcome measures will be assessed by blinded examiners at baseline and 12 weeks.

Chiropractic investigators from Northwestern Health Sciences University are collaborating with medical clinicians from the University of Minnesota, the Minneapolis Medical Research Foundation, and the Pain Assessment and Rehabilitation Center. This established team of investigators will work together in all phases of this innovative study, leading to dissemination and publication of study results and hypothesis generation for future research. This trial will yield important information allowing health care practitioners, policy makers and patients to make better-informed decisions regarding treatment choices for chronic neck pain. Importantly, it will serve to increase the extremely limited research that currently exists for this significant health-care condition.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical neck pain (defined as current episode > 12 weeks' duration).
* Quebec Task Force classifications 1, 2, 3 and 4. This includes patients with neck pain, stiffness or tenderness, with or without musculoskeletal and neurological signs.

Exclusion Criteria:

* Previous cervical spine surgery
* Neck pain referred from local joint lesions of the lower extremities or from visceral diseases
* Progressive neurological deficits due to nerve root or spinal cord compression
* Existing cardiac disease requiring medical treatment
* Blood clotting disorders
* Diffuse idiopathic hyperostosis
* Infectious and non-infectious inflammatory or destructive tissue changes of the cervical spine
* Presence of significant infectious disease, or other severe disabling health problems
* Substance abuse
* Ongoing treatment for neck pain by other health care providers
* Pregnant or nursing women
* Average neck pain score of less than 30 percentage points
* Pending or current litigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2001-03; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Patient rated pain(0-10 scale,11 box) | short term = 12 weeks; long term = 52 weeks

SECONDARY OUTCOMES:
Neck Disability Index (NDI)at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
General health status at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Improvement (Global Change)at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Disability Days at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Bothersomeness of Symptoms at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Frequency of Symptoms at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Patient Satisfaction at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Depression at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Medication use at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Fear-Avoidance Beliefs at baseline, weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
Cervical range of motion at baseline, weeks 4,12 | short term = 12 weeks
Cervical Strength and Endurance at baseline, weeks 4,12 | short term = 12 weeks
Health Care Costs and Utilization at weeks 4,12,26,52 | short term = 12 weeks; long term = 52 weeks
In-depth Interview at week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (1):
- Wolfe-Harris Center for Clinical Studies, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Evans R, Bronfort G, Schulz C, Maiers M, Bracha Y, Svendsen K, Grimm R, Garvey T, Transfeldt E. Supervised exercise with and without spinal manipulation performs similarly and better than home exercise for chronic neck pain: a randomized controlled trial. Spine (Phila Pa 1976). 2012 May 15;37(11):903-14. doi: 10.1097/BRS.0b013e31823b3bdf. PMID 22024905
- See also: Related Info — http://www.nwhealth.edu/research/WHCCS/